CLINICAL TRIAL: NCT05680987
Title: Utilizing the Retrograde Femoral Nail-Advanced for Fixation of Distal Femur and Femoral Shaft Fractures: A Prospective Case Series
Brief Title: Retrograde Femoral Nail-Advanced Outcomes for Fixation of Distal Femur and Femoral Shaft Fractures
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: DePuy Synthes (Industry)
Responsible Party: Principal Investigator, William Kent, Assistant Professor of Orthopaedic Surgery, University of California, San Diego
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 210669
Record Dates: First submitted 2022-12-19; First posted 2023-01-11 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Femoral Fracture
MeSH Terms: conditions — Femoral Fractures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Retrograde Femoral Nail-Advanced (Other)
  Interventions: Procedure: RFN-Advanced Retrograde Femoral Nailing System

INTERVENTIONS:
Procedure: RFN-Advanced Retrograde Femoral Nailing System — RFN-Advanced Retrograde Femoral Nailing System for patients with a distal femur or femoral shaft fracture requiring surgery

SUMMARY:
This project consists of a prospective and retrospective case series design. Study candidates will include all patients 18 years or older, who were evaluated at UCSD and found to have a distal femur or femoral shaft fracture requiring surgical fixation. Patients who consent to study participation will recieve the RFN-advanced Retrograde Femoral Nailing System implant for fracture fixation. Data on functional status, healing rates, complication rates, and pain levels will be collected for each participant. After 3 years of data collection, investigators will analyze this data to provide further insight on the utility of this new design of retrograde femoral nails. Given the relatively high rate of complications, such as malalignment, with current femoral nail designs, it is imperative to evaluate novel systems to appropriately manage distal femur or femoral shaft fractures.

ELIGIBILITY:
Inclusion Criteria:

* Distal femur or femoral shaft fracture requiring surgery
* Evaluation and treatment at UCSD
* Age 18 years or older
* Ability to understand the content of the patient information/Informed Consent Form
* Signed and dated IRB-approved written informed consent

Exclusion Criteria:

* Any not medically managed severe systemic disease
* their doctor has decided that it is in the patient's best interest to receive a different method of fixation
* Their doctor has determined that the patient has a condition that would make them unsuitable for participation in the study
* Pregnancy or women planning to conceive within the subject participation period (1 year) note: pregnancy will be self-reported and no test will be performed to test for it
* Prisoner
* Participation in any other pharmacologic or medicinal product study within the previous month that could influence the results of this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-06-23 (Actual); Primary Completion 2026-06-23 (Estimated); Study Completion 2026-06-23 (Estimated)

PRIMARY OUTCOMES:
Healing Rates | 2 years

SECONDARY OUTCOMES:
Pain Score (0-10,0=no pain, 10=most severe) | 1 year
Number of Complications | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- University of California, San Diego, San Diego, California, United States